CLINICAL TRIAL: NCT00306202
Title: Phase I Study of SRC/ABL Tyrosine Kinase Inhibitor Dasatinib [BMS-354825] in Children and Adolescents With Relapsed or Refractory Leukemia, Protocol ITCC 005
Brief Title: Study of Dasatinib in Children and Adolescents With Relapsed or Refractory Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Innovative Therapies For Children with Cancer Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-018; Protocol ITCC 005; 2005-002882-35 (EudraCT Number)
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Results first posted 2012-07-23 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Leukemia
Keywords: Relapsed and Refractory Leukemia
MeSH Terms: conditions — Leukemia; Recurrence | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stratum 1 (Ph+ CP-CML) (Experimental): Participants with imatinib-resistant Philadelphia chromosome positive (Ph+) chronic myeloid leukemia (CML) in chronic phase (CP)
  Interventions: Drug: Dasatinib
- Stratum 2/3 (Ph+ ALL or AP/BP-CML) (Experimental): Participants with imatinib-resistant or imatinib-intolerant Ph+ CML in accelerated phase (AP), or in myeloid blast phase (MBP), or in lymphoid blast phase (LBP); or relapsed or refractory Ph+ acute lymphoblastic leukemia (ALL) after imatinib use; or second or subsequent relapse of Ph+ acute myeloid leukemia (AML)
  Interventions: Drug: Dasatinib
- Stratum 4 (Ph- ALL/AML) (Experimental): Participants with second or subsequent relapse of Ph- ALL or Ph- AML
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, If necessary in participants who could not swallow, tablets were dispersed into 30 cc of 100% fruit juice with no preservatives (minute maid lemonade or orange juice or apple juice). Starting Dose Level of 60 mg/m^2; Escalated/Dose Level 2 of 80 mg/m^2. Once daily (QD), as long as clinical benefit was maintained.
  Intra-participant dose escalation was allowed based on tolerance and on individual response. The starting dose for subsequent participants in a stratum may have been escalated depending on safety, assessed by prior intra-participant dose-escalation, and lack of efficacy in previous participants. Treatment courses were defined as 3 weeks (21 days plus any required delay); for participants who stayed on treatment > 12 months, courses after 12 months were defined in quartiles of 13 weeks. Participants were to be followed until death or up to 5 years after end-of-treatment (EOT).
  Other Names: Sprycel; BMS-354825
  Arms: Stratum 1 (Ph+ CP-CML)
Drug: Dasatinib — Tablets, Oral, If necessary in participants who could not swallow, tablets were dispersed into 30 cc of 100% fruit juice with no preservatives (minute maid lemonade or orange juice or apple juice). Starting Dose Level of 60 mg/m^2; Escalated/Dose Level 2 of 80 mg/m^2. QD, as long as clinical benefit was maintained.
  Intra-participant dose escalation was allowed based on tolerance and on individual response. The starting dose for subsequent participants in a stratum may have been escalated depending on safety, assessed by prior intra-participant dose-escalation, and lack of efficacy in previous participants. Treatment courses were defined as 3 weeks (21 days plus any required delay); for participants who stayed on treatment > 12 months, courses after 12 months were defined in quartiles of 13 weeks. Participants were to be followed until death or up to 5 years after EOT.
  Other Names: Sprycel; BMS-354825
  Arms: Stratum 2/3 (Ph+ ALL or AP/BP-CML)
Drug: Dasatinib — Tablets, Oral, If necessary in participants who could not swallow, tablets were dispersed into 30 cc of 100% fruit juice with no preservatives (minute maid lemonade or orange juice or apple juice). Starting Dose Level of 60 mg/m^2; Escalated/Dose level 2 of 80 mg/m^2, Escalated/Dose level 3 of 100 mg/m^2, and Escalated/Dose level 4 of 120 mg/m^2. QD, as long as clinical benefit was maintained.
  Intra-participant dose escalation was allowed based on tolerance and on individual response. The starting dose for subsequent participants in a stratum may have been escalated depending on safety, assessed by prior intra-participant dose-escalation, and lack of efficacy in previous participants. Treatment courses were defined as 3 weeks (21 days plus any required delay); for participants who stayed on treatment > 12 months, courses after 12 months were defined in quartiles of 13 weeks. Participants were to be followed until death or up to 5 years after EOT.
  Other Names: Sprycel; BMS-354825
  Arms: Stratum 4 (Ph- ALL/AML)

SUMMARY:
The purpose of this clinical research study was to establish a recommended phase 2 once daily (QD) dose of dasatinib and to assess the efficacy of the investigational drug for relapsed or refractory (resistant to previous treatment) leukemia in children and adolescents. The side effects that this oral investigational drug may have in children, and the levels of the drug in the blood, will be studied at different doses.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Ph-positive (Ph+) Chronic Myelogenous Leukemia in chronic, accelerated or blast phase or Ph+ acute lymphoblastic leukemia (ALL) with imatinib-resistant disease or intolerance to imatinib.
* Ph-negative acute leukemia in second or subsequent relapse
* Age >1 and <21 years
* Lansky or Karnofsky scale >60
* Life expectancy >3 weeks
* Adequate hepatic and renal function
* Written informed consent

Exclusion Criteria:

* Subjects for whom potentially-curative therapy was available, including electing immediate [ie, planned <45 days] stem-cell transplantation. Subjects in Stratum 1 were to have had an ongoing identical HLA donor search, and may have discontinued study if a donor became available.)
* Subjects with symptomatic central nervous system (CNS) disease (eg, convulsions due to their CNS disease).
* Subjects who had not recovered from acute toxicity of previous therapy.
* Clinically-significant disorder of platelet function (eg, von Willebrand's disease) or ongoing gastrointestinal bleeding.
* Serious uncontrolled medical disorder or active infection
* Uncontrolled or significant cardiovascular disease
* Use of any investigational agent or any other anticancer agent within 14 days prior to treatment start.
* Prior therapy with dasatinib
* Subjects taking medications that irreversibly inhibit platelet function or anticoagulants.
* Subjects taking certain medications that are accepted to have a risk of causing QTc prolongation.
* Women of Child Bearing Potential with a positive pregnancy test prior to study drug administration.
* Expected noncompliance, or unable to have regular follow-up due to psychologic, social, familial, or geographic reasons.
* Subjects who are compulsorily detained for legal reasons or treatment of either a psychiatric or physical (eg, infectious disease) illness must not be enrolled into this study.

Ages: 12 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2006-03-31 (Actual); Primary Completion 2011-05-31 (Actual); Study Completion 2019-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- Local Institution, Vienna, Austria
- France (2):
  - Local Institution, Nantes
  - Local Institution, Paris
- Germany (3):
  - Local Institution, Berlin
  - Local Institution, Frankfurt
  - Local Institution, Hanover
- Local Institution, Monza (mi), Italy
- Local Institution, Rotterdam, Netherlands
- United Kingdom (4):
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Bristol, Somerset
  - Local Institution, Sutton, Surrey
  - Local Institution, Birmingham, West Midlands

REFERENCES:
- [Derived] Zwaan CM, Rizzari C, Mechinaud F, Lancaster DL, Lehrnbecher T, van der Velden VH, Beverloo BB, den Boer ML, Pieters R, Reinhardt D, Dworzak M, Rosenberg J, Manos G, Agrawal S, Strauss L, Baruchel A, Kearns PR. Dasatinib in children and adolescents with relapsed or refractory leukemia: results of the CA180-018 phase I dose-escalation study of the Innovative Therapies for Children with Cancer Consortium. J Clin Oncol. 2013 Jul 1;31(19):2460-8. doi: 10.1200/JCO.2012.46.8280. Epub 2013 May 28. PMID 23715577
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose: Participants with imatinib-resistant Philadelphia chromosome positive (Ph+) chronic myeloid leukemia (CML) in chronic phase (CP). Starting Dose Level of 60 mg/m^2; Escalated/Dose Level 2 of 80 mg/m^2. Once daily (QD), as long as clinical benefit was maintained.
- Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose: Participants with imatinib-resistant or imatinib-intolerant Ph+ CML in accelerated phase (AP), or in myeloid blast phase (MBP), or in lymphoid blast phase (LBP); or relapsed or refractory Ph+ acute lymphoblastic leukemia (ALL) after imatinib use; or second or subsequent relapse of Ph+ acute myeloid leukemia (AML). Starting Dose Level of 60 mg/m^2; Escalated/Dose level 2 of 80 mg/m^2. QD, as long as clinical benefit was maintained.
- Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose: Participants with second or subsequent relapse of Ph- ALL or Ph- AML. Starting Dose Level of 60 mg/m^2; Escalated/Dose level 2 of 80 mg/m^2, Escalated/Dose level 3 of 100 mg/m^2, and Escalated/Dose level 4 of 120 mg/m^2. QD, as long as clinical benefit was maintained.
Period: Overall Study
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose | Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose
Started | 17 (Started = Treated. 18 were enrolled; 1 no longer met study criteria and was never treated) | 17 (Started=Treated. 20 were enrolled;3 never treated(2 no longer met study criteria;1 withdrew consent)) | 24 (Started = Treated. 25 were enrolled; 1 no longer met study criteria and was never treated)
Completed | 17 (Completed = Off-treatment) | 17 (Completed = Off-treatment) | 24 (Completed = Off-treatment)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose | Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose | Total
Number analyzed (Participants) | 17 | 17 | 24 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (4.1) | 9.7 (4.3) | 8.6 (5.6) | 10.0 (5.0)
Age, Customized [Number; unit: Participants]
  < 2 years | 0 | 0 | 2 | 2
  Between 2 and 6 years | 2 | 5 | 7 | 14
  Between 7 and 11 years | 6 | 5 | 7 | 18
  Between 12 and 18 years | 9 | 7 | 7 | 23
  > 18 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 8 | 19
  Male | 11 | 12 | 16 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 0 | 1
  Unknown or Not Reported | 17 | 16 | 24 | 57
Race/Ethnicity, Customized [Number; unit: Participants] — Race only
  Participants
    White | 16 | 15 | 21 | 52
    Black/African American | 0 | 0 | 1 | 1
    Asian | 1 | 1 | 1 | 3
    Other | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose of Dasatinib in Children and Adolescents With Relapsed or Refractory Leukemia
Description: The recommended phase 2 dasatinib dose was determined based on efficacy, safety, and pharmacokinetic data obtained at the prespecified dose levels.
Time Frame: From the date of first dose to end-of-treatment (EOT) (Median duration of therapy in months: Stratum 1=24.11 [Range:2.27-50.63]; Stratum 2/3=3.02 [Range: 0.53-37.72]; Stratum 4=1.14 [Range: 0.03-3.38])
Population: All treated participants: Participants who received at least 1 dose of study therapy
Measure: Number; unit: mg/m^2 QD
Groups:
- Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose: Participants with second or subsequent relapse of Ph- ALL or Ph- AML. Starting Dose Level of 60 mg/m^2; Escalated/Dose Level 2 of 80 mg/m^2, escalated/dose level 3 of 100 mg/m^2, escalated/dose level 3 of 120 mg/m^2. QD, as long as clinical benefit was maintained.
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose | Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose
Number analyzed (Participants) | 17 | 17 | 24
mg/m^2 QD | 60 | 80 | NA — Phase II dose was not chosen for this population as there is no current plan to move forward with development in this population due to lack of efficacy despite escalations to the highest dose of 120 mg/m^2 in this trial.

2. Secondary Outcome: Number of Participants With Related Deaths, Serious Adverse Events (SAEs), and Adverse Events (AEs) by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0.
Description: AE: New untoward medical occurrence or worsening of a preexisting medical condition that does not have causal relationship with this treatment. SAE: Untoward medical event that at any dose: results in death, persistent or significant disability/incapacity, drug dependency/abuse; life-threatening, an important medical event, a congenital anomaly/birth defect; requires inpatient hospitalization/prolongs existing hospitalization. Grade 3 = Severe; Grade 4 = Life-threatening or disabling.
Time Frame: From the date of first dose until at least 30 days after the last dose of study drug (Median duration of therapy in months: Stratum 1=24.11 [Range: 2.27-50.63]; Stratum 2/3=3.02 [Range: 0.53-37.72]; Stratum 4=1.14 [Range: 0.03-3.38])
Population: All treated participants: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Groups:
- Stratum 1 Ph+ CP-CML (Dasatinib 60 mg/m^2): Participants with imatinib-resistant Philadelphia chromosome positive (Ph+) chronic myeloid leukemia (CML) in chronic phase (CP). Dasatinib 60 mg/m^2 QD, as long as clinical benefit was maintained.
- Stratum 1 Ph+ CP-CML (Dasatinib 80 mg/m^2): Participants with imatinib-resistant Philadelphia chromosome positive (Ph+) chronic myeloid leukemia (CML) in chronic phase (CP). Dasatinib 80 mg/m^2 QD, as long as clinical benefit was maintained.
- Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 60 mg/m^2): Participants with imatinib-resistant or imatinib-intolerant Ph+ CML in accelerated phase (AP), or in myeloid blast phase (MBP), or in lymphoid blast phase (LBP); or relapsed or refractory Ph+ acute lymphoblastic leukemia (ALL) after imatinib use; or second or subsequent relapse of Ph+ acute myeloid leukemia (AML). Dasatinib 60 mg/m^2 QD, as long as clinical benefit was maintained.
- Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 80 mg/m^2): Participants with imatinib-resistant or imatinib-intolerant Ph+ CML in accelerated phase (AP), or in myeloid blast phase (MBP), or in lymphoid blast phase (LBP); or relapsed or refractory Ph+ acute lymphoblastic leukemia (ALL) after imatinib use; or second or subsequent relapse of Ph+ acute myeloid leukemia (AML). Dasatinib 80 mg/m^2 QD, as long as clinical benefit was maintained.
- Stratum 4 Ph- ALL/AML (Dasatinib 60 mg/m^2): Participants with second or subsequent relapse of Ph- ALL or Ph- AML. Dasatinib 60 mg/m^2 QD, as long as clinical benefit was maintained.
- Stratum 4 Ph- ALL/AML (Dasatinib 80 mg/m^2): Participants with second or subsequent relapse of Ph- ALL or Ph- AML. Dasatinib 80 mg/m^2 QD, as long as clinical benefit was maintained.
- Stratum 4 Ph- ALL/AML (Dasatinib 100 mg/m^2): Participants with second or subsequent relapse of Ph- ALL or Ph- AML. Dasatinib 100 mg/m^2 QD, as long as clinical benefit was maintained.
- Stratum 4 Ph- ALL/AML (Dasatinib 120 mg/m^2): Participants with second or subsequent relapse of Ph- ALL or Ph- AML. Dasatinib 120 mg/m^2 QD, as long as clinical benefit was maintained.
Arm/Group | Stratum 1 Ph+ CP-CML (Dasatinib 60 mg/m^2) | Stratum 1 Ph+ CP-CML (Dasatinib 80 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 60 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 80 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 60 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 80 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 100 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 120 mg/m^2)
Number analyzed (Participants) | 11 | 6 | 8 | 9 | 6 | 6 | 6 | 6
participants
  Drug-Related Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Drug-Related SAEs | 1 | 1 | 2 | 3 | 2 | 2 | 2 | 2
  Drug-Related AEs Leading to Discontinuation | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Grade 3/4 AEs | 5 | 3 | 4 | 3 | 3 | 4 | 3 | 2

3. Secondary Outcome: Number of Participants With Dose-limiting Toxicity (DLT)
Description: DLTs: AEs which were at least possibly drug-related occurring within first 3 weeks of dasatinib therapy (toxicities occurring after 21 days were also considered) and are:- --Any nonhematologic clinically-apparent toxicity of Grade(GR)≥3 occurring despite appropriate medical management and GR4 laboratory abnormality/GR3 lasting ≥7 days --GR4 neutropenia or thrombocytopenia lasting ≥7 days and not explained by the presence of leukemia after hematopoietic reconstitution --Any clinically important toxicity of GR≥2 requiring treatment discontinuation or interruption ≥7 days.
Time Frame: as for outcome 2
Population: All treated participants: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum 1 Ph+ CP-CML (Dasatinib 60 mg/m^2) | Stratum 1 Ph+ CP-CML (Dasatinib 80 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 60 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 80 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 60 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 80 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 100 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 120 mg/m^2)
Number analyzed (Participants) | 11 | 6 | 8 | 9 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

4. Secondary Outcome: Number of Participants With Hematology Abnormalities by NCI CTCAE Version 3.0
Description: GR1=Mild; GR2=Moderate; GR3=Severe; GR4=Life-threatening or disabling. Normal ranges provided by local laboratory and may also vary from site to site. WBC: GR1=<LLN-3.0*10^9/L; GR2=<3.0-2.0*10^9/L; GR3=<2.0-1.0*10^9/L; GR4=<1.0*10^9/L. ANC: GR1=<LLN-1.5*10^9 /L; GR2=<1.5-1.0*10^9/L; GR3=<1.0-0.5*10^9/L; GR4=<0.5*10^9/L. Hemoglobin: GR1=<LLN-10.0g/dL; GR2=<10.0-8.0g/dL; GR3=<8.0-6.5g/dL; GR4=<6.5g/dL. Platelets: GR1=<LLN-75.0*10^9/L; GR2=<75.0-50.0*10^9/L; GR3=<50.0-25.0*10^9/L; GR4=<25.0*10^9/L.
Time Frame: Days 8, 15, 22, 29, 36, 43, then every 3 weeks, then every 3 months after 1 Year, EOT (Median duration of therapy in months: Stratum 1=24.11 [Range: 2.27-50.63]; Stratum 2/3=3.02 [Range: 0.53-37.72]; Stratum 4=1.14 [Range: 0.03-3.38])
Population: All treated participants: Participants who received at least one dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum 1 Ph+ CP-CML (Dasatinib 60 mg/m^2) | Stratum 1 Ph+ CP-CML (Dasatinib 80 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 60 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 80 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 60 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 80 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 100 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 120 mg/m^2)
Number analyzed (Participants) | 11 | 6 | 8 | 9 | 6 | 6 | 6 | 6
participants
  WBC GR1 | 6 | 4 | 2 | 1 | 1 | 1 | 0 | 0
  WBC GR2 | 0 | 1 | 3 | 3 | 0 | 1 | 1 | 1
  WBC GR3 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
  WBC GR4 | 0 | 0 | 1 | 3 | 2 | 2 | 3 | 1
  ANC GR1 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0
  ANC GR2 | 4 | 0 | 2 | 2 | 1 | 0 | 0 | 0
  ANC GR3 | 1 | 2 | 2 | 0 | 0 | 2 | 0 | 2
  ANC GR4 | 0 | 1 | 3 | 4 | 4 | 4 | 6 | 3
  Platelet GR1 | 4 | 4 | 0 | 2 | 0 | 0 | 0 | 0
  Platelet GR2 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0
  Platelet GR3 | 2 | 0 | 4 | 1 | 0 | 1 | 1 | 1
  Platelet GR4 | 0 | 0 | 4 | 3 | 4 | 5 | 5 | 5
  Hemoglobin GR1 | 3 | 4 | 1 | 0 | 0 | 0 | 0 | 0
  Hemoglobin GR2 | 4 | 1 | 5 | 3 | 2 | 3 | 3 | 3
  Hemoglobin GR3 | 0 | 0 | 1 | 4 | 3 | 1 | 3 | 2
  Hemoglobin GR4 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0

5. Secondary Outcome: Number of Participants With Serum Chemistry Abnormalities (Calcium, Magnesium, and Phosphate) by NCI CTCAE Version 3.0
Description: GR1=Mild; GR2=Moderate; GR3=Severe; GR4=Life-threatening or disabling. Normal ranges provided by local laboratory and may also vary from site to site. Low calcium: GR1=<LLN-8.0 mg/dL, GR2=<8.0-7.0 mg/dL, GR3=<7.0-6.0 mg/dL, GR4=<6.0 mg/dL; Low magnesium: GR1=<LLN-1.2 mg/dL, GR2=<1.2-0.9 mg/dL, GR3=<0.9-0.7 mg/dL, GR4=<0.7 mg/dL; Low phosphate: GR1=<LLN - 2.5 mg/dL, GR2=<2.5 - 2.0 mg/dL, GR3=<2.0 - 1.0 mg/dL, GR4=<1.0 mg/dL.
Time Frame: Days 22 and 43, then every 12 weeks, then every 24 weeks after 24 months of treatment, EOT (Median duration of therapy in months: Stratum 1=24.11 [Range: 2.27-50.63]; Stratum 2/3=3.02 [Range: 0.53-37.72]; Stratum 4=1.14 [Range: 0.03-3.38])
Population: All treated participants: Participants who received at least one dose of study therapy.
Measure: Number; unit: participants
Groups:
- Stratum 1 Ph+ CP-CML (Dasatinib 80 mg/m^2): Participants with imatinib-resistant Philadelphia chromosome positive (Ph+) chronic myeloid leukemia (CML) in chronic phase (CP). Dasatinib 80 mg/m^2, as long as clinical benefit was maintained.
Arm/Group | Stratum 1 Ph+ CP-CML (Dasatinib 60 mg/m^2) | Stratum 1 Ph+ CP-CML (Dasatinib 80 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 60 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 80 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 60 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 80 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 100 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 120 mg/m^2)
Number analyzed (Participants) | 11 | 6 | 8 | 9 | 6 | 6 | 6 | 6
participants
  Low Calcium GR1 | 3 | 0 | 2 | 2 | 2 | 0 | 1 | 0
  Low Calcium GR2 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 1
  Low Calcium GR3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Low Calcium GR4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Low magnesium GR1 | 1 | 1 | 5 | 0 | 1 | 0 | 4 | 1
  Low Magnesium GR2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Low Magnesium GR3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Low Magnesium GR4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Low Phosphate GR1 | 2 | 1 | 2 | 2 | 0 | 2 | 2 | 1
  Low Phosphate GR2 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1
  Low Phosphate GR3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  Low Phosphate GR4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Serum Chemistry Abnormalities (Liver and Renal Function) by NCI CTCAE Version 3.0
Description: GR1=Mild; GR2=Moderate; GR3=Severe; GR4=Life-threatening or disabling. Normal ranges provided by local laboratory and may also vary from site to site. AST and ALT: GR1=>ULN-2.5*ULN; GR2=>2.5-5.0*ULN; GR3=>5.0-20.0*ULN; GR4:>20.0*ULN. Total bilirubin:GR1=>ULN-1.5*ULN, GR2=>1.5-3.0*ULN, GR3=>3-10*ULN, GR4=>10*ULN. Creatinine: GR1=>ULN-1.5*ULN, GR2=>1.5-3.0*ULN, GR3=>3.0-6.0*ULN, GR4=>6.0*ULN.
Time Frame: as for outcome 5
Population: All treated participants: Participants who received at least one dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum 1 Ph+ CP-CML (Dasatinib 60 mg/m^2) | Stratum 1 Ph+ CP-CML (Dasatinib 80 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 60 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 80 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 60 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 80 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 100 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 120 mg/m^2)
Number analyzed (Participants) | 11 | 6 | 8 | 9 | 6 | 6 | 6 | 6
participants
  AST GR1 | 1 | 3 | 5 | 3 | 1 | 4 | 2 | 2
  AST GR2 | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 1
  AST GR3 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0
  AST GR4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  High ALT GR1 | 4 | 4 | 4 | 2 | 0 | 2 | 3 | 2
  High ALT GR2 | 0 | 0 | 2 | 1 | 1 | 2 | 1 | 0
  High ALT GR3 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1
  High ALT GR4 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Total Bilirubin GR1 | 2 | 0 | 1 | 1 | 0 | 1 | 2 | 0
  Total Bilirubin GR2 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1
  Total Bilirubin GR3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin GR4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  High Serum Creatinine GR1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0
  High Serum Creatinine GR2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  High Serum Creatinine GR3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  High Serum Creatinine GR4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Major Cytogenetic Response (MCyR) at Any Time in Stratum 1 (Ph+ CP-CML) and Stratum 2/3 (Ph+ ALL or AP/BP-CML)
Description: Cytogenetic responses were based on the karyotype analysis of the percentage of Ph+ metaphases among cells in metaphase on a BM sample. At least 20 metaphase cells from a BM sample were evaluated. MCyR: A cytogenetic response that is either complete cytogenetic response (CCyR) or partial cytogenetic response (PCyR). CCyR: 0% Ph+ cells in metaphase in BM. PCyR: >0% to 35% Ph+ cells in metaphase in BM.
Time Frame: Strata 1 and 2/3: At Week 7, 13, then every 12 weeks, and EOT; Stratum 2/3: Additionally at Week 4, 19, 31 (Median duration of therapy in months: Stratum 1=24.11 [Range: 2.27-50.63]; Stratum 2/3=3.02 [Range: 0.53-37.72])
Population: All treated participants in strata 1 and 2/3: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Groups:
- Stratum 1 Ph+ CP-CML (Dasatinib 80 mg/m^2): Participants with imatinib-resistant Ph+ chronic myeloid leukemia (CML) in chronic phase (CP). Dasatinib 80 mg/m^2 QD, as long as clinical benefit was maintained.
Arm/Group | Stratum 1 Ph+ CP-CML (Dasatinib 60 mg/m^2) | Stratum 1 Ph+ CP-CML (Dasatinib 80 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 60 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 80 mg/m^2)
Number analyzed (Participants) | 11 | 6 | 8 | 9
participants | 9 | 6 | 4 | 7

8. Secondary Outcome: Number of Participants With Major Cytogenetic Response (MCyR) in Stratum 1 (Ph+ CP-CML) Within First 12 and 24 Weeks
Description: Cytogenetic responses were based on the karyotype analysis of the percentage of Ph+ metaphases among cells in metaphase on a BM sample. At least 20 metaphase cells from a BM sample were evaluated. MCyR: A cytogenetic response that was either CCyR or PCyR. CCyR: 0% Ph+ cells in metaphase in BM. PCyR: >0% to 35% Ph+ cells in metaphase in BM.
Time Frame: After completion of Week 12 and 24 (measured at Weeks 13 and 25)
Population: All treated participants in stratum 1: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum 1 Ph+ CP-CML (Dasatinib 60 mg/m^2) | Stratum 1 Ph+ CP-CML (Dasatinib 80 mg/m^2)
Number analyzed (Participants) | 11 | 6
participants
  MCyR within first 12 weeks | 6 | 2
  MCyR within first 24 weeks | 9 | 5

9. Secondary Outcome: Best Cytogenetic Response (CyR) in Stratum 1 (Ph+ CP-CML) and Stratum 2/3 (Ph+ ALL or AP/BP-CML)
Description: Best CyR was assessed based on the percentages of Ph+ metaphases of ≥20 analyzed metaphases in BM sample. Participants with complete, partial, minor, minimal, or no CyR. Refer to Outcome Measure 7 for definitions of CCyR and PCyR. Minor CyR:>35%-65% Ph+ cells in metaphase in BM. Minimal CyR:>65%-95% Ph+ cells in metaphase in BM. No CyR:>95%-100% Ph+ cells in metaphase in BM. Unable to determine:Participants without valid cytogenetic assessment (i.e., at least 1 metaphase observed and number of Ph+ metaphases smaller than total number of metaphases [%Ph+ <100%]).
Time Frame: Strata 1 and 2/3: At Weeks 7, 13, then every 12 weeks, and EOT; Stratum 2/3: Additionally at Weeks 4, 19, 25, 31 (Median duration of therapy in months: Stratum 1=24.11 [Range: 2.27-50.63]; Stratum 2/3=3.02 [Range: 0.53-37.72])
Population: All treated participants (strata 1 and 2/3): Participants who received at least 1 dose of study therapy. Stratum 2/3 dasatinib 80 mg/m^2 dose cohort includes 1 participant as having a CCyR due to a data entry error that was fixed after database lock for this study.
Measure: Number; unit: participants
Arm/Group | Stratum 1 Ph+ CP-CML (Dasatinib 60 mg/m^2) | Stratum 1 Ph+ CP-CML (Dasatinib 80 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 60 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 80 mg/m^2)
Number analyzed (Participants) | 11 | 6 | 8 | 9
participants
  No Response (>95% - 100%) | 1 | 0 | 0 | 1
  Minimal (>65% - 95%) | 0 | 0 | 0 | 0
  Minor (>35% - 65%) | 1 | 0 | 0 | 0
  Partial (>0% - 35%) | 1 | 0 | 0 | 0
  Complete (0%) | 8 | 6 | 4 | 8
  Unable to determine | 0 | 0 | 4 | 0

10. Secondary Outcome: Percentage of Participants With Complete Cytogenetic Response (CCyR) or Major Cytogenetic Response (MCyR) at Recommended Phase II Dose
Description: as for outcome 8
Time Frame: as for outcome 7
Population: All treated participants in strata 1 and 2/3: Participants who received at least 1 dose of study therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1 Ph+ CP-CML (Dasatinib 60 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 80 mg/m^2)
Number analyzed (Participants) | 11 | 9
percentage of participants
  CCyR | 72.7 [39.0 to 94.0] | 88.9 [51.8 to 99.7]
  MCyR | 81.8 [48.2 to 97.7] | 88.9 [51.8 to 99.7]

11. Secondary Outcome: Time to Major Cytogenetic Response (MCyR) in Responders: Stratum 1 (Ph+ CP-CML) and Stratum 2/3 (Ph+ ALL or AP/BP-CML)
Description: Defined as time (in days) from the first dose of dasatinib until criteria were first met for MCyR. MCyR: A CyR that was either CCyR or PCyR. CCyR: 0% Ph+ cells in metaphase in BM. PCyR: >0% to 35% Ph+ cells in metaphase in BM. The Kaplan-Meier plot was used. A 2-sided, 95% confidence interval (CI) for the median was computed using the Brookmeyer and Crowley method.
Time Frame: Strata 1 and 2/3: At Weeks 7, 13, 25, 37, then every 12 weeks; Stratum 2/3: Additionally at Weeks 4, 19, 31; until first MCyR (maximum participant time to first MCyR of 92 days).
Population: All treated participants who had cytogenetic response. Participants with at least 1 metaphase observed & the number of Ph+ metaphases smaller than the total number of metaphases [%Ph+ <100%]) were considered responders.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose: Participants with imatinib-resistant Philadelphia chromosome positive (Ph+) chronic myeloid leukemia (CML) in chronic phase (CP). Starting Dose Level of 60 mg/m^2; Escalated/Dose level 2 of 80 mg/m^2. QD, as long as clinical benefit was maintained.
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose
Number analyzed (Participants) | 15 | 12
days | 75.0 [43.0 to 92.0] | 33.5 [22.0 to 43.0]

12. Secondary Outcome: Duration of Major Cytogenetic Response (MCyR) in Responders (Stratum 1 [Ph+ CP-CML] and Stratum 2/3 [Ph+ ALL or AP/BP-CML])
Description: Defined as the time (in months) from the first day that all criteria were met for MCyR until the date of progression (based on the Investigator's assessment) or death (for participants whose best responses were MCyR and CCyR respectively). MCyR: A cytogenetic response that was either CCyR or PCyR. CCyR: 0% Ph+ cells in metaphase in BM. PCyR: >0% to 35% Ph+ cells in metaphase in BM. The Kaplan-Meier plot was used. A 2-sided, 95% CI for the median was computed using the Brookmeyer and Crowley method.
Time Frame: From the date of first MCyR assessment to date of progression, death, or last tumor assessment (maximum participant duration of response of 48.6 months)
Population: All treated participants who had cytogenetic response. Participants with at least 1 metaphase observed & the number of Ph+ metaphases smaller than the total number of metaphases [%Ph+ <100%]) were considered responders. Participants who neither progressed nor died were censored on the date of their last valid cytogenetic assessment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose: Participants with imatinib-resistant Philadelphia chromosome positive (Ph+) chronic myeloid leukemia (CML) in chronic phase (CP). Starting Dose Level of 60 mg/m^2; Escalated/Dose level 1 of 80 mg/m^2. QD, as long as clinical benefit was maintained.
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose
Number analyzed (Participants) | 15 | 12
months | 52.2 [10.0 to 56.1] | 4.6 [1.2 to 17.4]

13. Secondary Outcome: Duration of Complete Cytogenetic Response (CCyR) in Responders: Stratum 1 [Ph+ CP-CML] and Stratum 2/3 [Ph+ ALL or AP/BP-CML]
Description: Defined as time (in months) from the first day that all criteria were met for CCyR until the date of progression (based on the Investigator's assessment) or death (for participants whose best response was CCyR). CCyR = 0% Ph+ metaphases of ≥ 20 analyzed metaphases in BM aspiration. The Kaplan-Meier plot was used. A 2-sided, 95% CI for the median was computed using the Brookmeyer and Crowley method.
Time Frame: From the date of first CCyR assessment to date of progression, death, or last tumor assessment (maximum participant duration of response of 45.1 months)
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose
Number analyzed (Participants) | 14 | 12
months | 48.1 [10.0 to 56.1] | 4.6 [1.2 to 17.4]

14. Secondary Outcome: Number of Participants With Major Hematologic Response (MaHR) at Any Time in Stratum 2/3 (Ph+ ALL or AP/BP-CML) and Stratum 4 (Ph- ALL/AML)
Description: Defined as participants having as best response complete hematologic response (CHR) or CHR with incomplete platelet recovery (CHRp). Criteria: CHR-WBC in Peripheral Blood (PB):≤ULN; Immature cells in PB:No blasts, promyelocytes, myelocytes, metamyelocytes; Platelet count (untransfused):≥100,000/mm^3 and ≤450,000/mm^3; ANC:≥ 1000/mm^3; Blasts in BM:<5%; Extra medullary disease:No extramedullary leukemia, including no hepato or splenomegaly (regardless of CNS involvement). CHRp-CHR except platelet count (untransfused) & ANC:20,000/mm^3 ≤platelet <100,000/mm^3 & /or 500/mm^3 ≤ANC ≤1000/mm^3.
Time Frame: Days 8, 15, 22, 29, 36, 43; Weeks 4, 7, 13, 19, 25, 31, 37; at Week 10 (only stratum 4); then every 12 weeks upto 24 months; then once/year; EOT(Median duration of therapy in months: Stratum 2/3=3.02 [Range: 0.53-37.72]; Stratum 4=1.14 [Range: 0.03-3.38])
Population: All treated participants in strata 2/3 and 4: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 60 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 80 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 60 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 80 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 100 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 120 mg/m^2)
Number analyzed (Participants) | 8 | 9 | 6 | 6 | 6 | 6
participants | 2 | 6 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Major Hematologic Response (MaHR) in Stratum 2/3 (Ph+ ALL or AP/BP-CML) Within First 6 and 24 Weeks
Description: Defined as participants having as best response a CHR or CHRp. Criteria: CHR-WBC in PB:≤ULN; Immature cells in PB:No blasts, promyelocytes, myelocytes, metamyelocytes; Platelet count (untransfused):≥100,000/mm^3 and ≤450,000/mm^3; ANC:≥ 1000/mm^3; Blasts in BM:<5%; Extra medullary disease:No extramedullary leukemia, including no hepato or splenomegaly (regardless of CNS involvement). CHRp-CHR except platelet count (untransfused) and ANC:20,000/mm^3 ≤platelet <100,000/mm^3 and /or 500/mm^3 ≤ANC ≤1000/mm^3.
Time Frame: After completion of Week 6 and 24 (measured at weeks 7 and 25)
Population: All treated participants in Stratum 2/3: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 60 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 80 mg/m^2)
Number analyzed (Participants) | 8 | 9
participants
  MaHR within first 6 weeks | 2 | 5
  MaHR within first 24 weeks | 2 | 6

16. Secondary Outcome: Best Hematologic Response (HR) At Any Time: Stratum 1 (Ph+ CP-CML)
Description: HR: Determined by complete blood count (CBC), differential, and platelet count (PLT). Criteria for complete hematologic response (CHR): WBC in PB: <10,000/mm^3; Immature cells in PB: No blasts or promyelocytes (myelocytes + metamyelocytes) <5%; Basophils in PB: <5%; Platelet count (untransfused): <450,000/mm^3; Extra medullary disease: No extramedullary leukemia, including no splenomegaly. Unconfirmed HR = All criteria met. Confirmed HR = Criteria for HR fulfilled again at least 28 days after they first met with no concomitant use of anagrelide or hydroxyurea during this interval.
Time Frame: Days 8, 15, 22, 29, 36, 43; Weeks 7, 13, 25, 37; then every 12 weeks upto 24 months; then once/year; EOT (Median duration of therapy in months: Stratum 1=24.11 [Range: 2.27-50.63])
Population: All treated participants in stratum 1: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum 1 Ph+ CP-CML (Dasatinib 60 mg/m^2) | Stratum 1 Ph+ CP-CML (Dasatinib 80 mg/m^2)
Number analyzed (Participants) | 11 | 6
participants
  Best Confirmed HR-Complete | 10 | 6
  Best Confirmed HR-No Response | 1 | 0
  Best Unconfirmed Hematologic Response-Complete | 10 | 6
  Best Unconfirmed Hematologic Response-No Response | 1 | 0

17. Secondary Outcome: Best Hematologic Response (HR) At Any Time: Stratum 2/3 (Ph+ ALL or AP/BP-CML)
Description: HR was determined by CBC, differential, and platelet count. Refer to outcome measure 15 for criteria for CHR and CHRp. Criteria for minor hematologic response (MiHR): CHRp except blasts in BM-≥5% and ≤15% blasts in BM. Unconfirmed HR = All criteria met. periph=peripheral. Confirmed HR = Criteria for HR fulfilled again at least 28 days after they first met with no concomitant use of anagrelide or hydroxyurea during this interval.
Time Frame: Days 8, 15, 22, 29, 36, 43; Weeks 4, 7, 13, 19, 25, 31, 37; then every 12 weeks up to 24 months; then once/year; EOT (Median duration of therapy in months: Stratum 2/3=3.02 [Range: 0.53-37.72])
Population: All treated participants in Stratum 2/3: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 60 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 80 mg/m^2)
Number analyzed (Participants) | 8 | 9
participants
  Best Confirmed HR-Complete | 1 | 5
  Best Confirmed HR-Complete except periph. recovery | 1 | 1
  Best Confirmed HR-No Response | 6 | 3
  Best Unconfirmed HR-Complete | 3 | 7
  Best Unconfirmed HR-Minor | 0 | 1
  Best Unconfirmed HR-No Response | 5 | 1

18. Secondary Outcome: Best Hematologic Response (HR) At Any Time: Stratum 4 (Ph- ALL/AML)
Description: HR was determined by CBC, differential, and platelet count. Unable to determine = Participants without any valid hematologic assessments.
Time Frame: Days 8, 15, 22, 29, 36, 43; Weeks 4, 7, 10, 13, 19, 25, 31, 37; then every 12 weeks upto 24 months; then once/year; EOT (Median duration of therapy in months: Stratum 4=1.14 [Range: 0.03-3.38])
Population: All treated participants in stratum 4: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum 4 Ph- ALL/AML (Dasatinib 60 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 80 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 100 mg/m^2) | Stratum 4 Ph- ALL/AML (Dasatinib 120 mg/m^2)
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants
  Best Confirmed HR-No Response | 5 | 6 | 6 | 6
  Best Confirmed HR-Unable to Determine | 1 | 0 | 0 | 0
  Best Unconfirmed HR-No Response | 5 | 6 | 6 | 6
  Best Unconfirmed HR-Unable to Determine | 1 | 0 | 0 | 0

19. Secondary Outcome: Time to Major Hematologic Response (MaHR): Stratum 2/3 (PH+ ALL or AP/BP-CML)
Description: Defined as time (in days) from first dose of dasatinib until the first day MaHR criteria were met, provided they were confirmed later (after 28 days) with no concomitant use of anagrelide or hydroxyurea during this interval. MaHR: Defined as participants having as best response a CHR or CHRp. Refer to Outcome Measure 15 for criteria for CHR and CHRp. Estimated by the Kaplan-Meier method and a 2-sided, 95% CI for the median was computed using the Brookmeyer and Crowley method.
Time Frame: Days 8, 15, 22, 29, 36, 43; Weeks 4, 7, 13, 19, 25, 31, 37; then every 12 weeks upto 24 months; then once/year; until confirmed MaHR (maximum participant time to first MaHR of 44 days).
Population: Treated participants with MaHR in stratum 2/3.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose: Participants with imatinib-resistant or imatinib-intolerant Ph+ CML in accelerated phase (AP), or in myeloid blast phase (MBP), or in lymphoid blast phase (LBP); or relapsed or refractory Ph+ acute lymphoblastic leukemia (ALL) after imatinib use; or second or subsequent relapse of Ph+ acute myeloid leukemia (AML). Starting Dose Level of 60 mg/m^2; Escalated/Dose level 2 of 80 mg/m^2 QD, as long as clinical benefit was maintained.
Arm/Group | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose
Number analyzed (Participants) | 8
days | 36.0 [29.0 to 42.0]

20. Secondary Outcome: Time to Complete Hematologic Response (CHR): Stratum 1 (Ph+ CP-CML) and Stratum 2/3 (Ph+ALL or AP/BP-CML)
Description: Time to CHR is the time (in days) from first dose of dasatinib until the first day CHR criteria were met, provided they were confirmed later after 28 days with no concomitant use of anagrelide or hydroxyurea during this interval. Refer to Outcome Measure 16 for criteria to CHR in Stratum 1 and to Outcome Measure 15 for criteria for CHR in Stratum 2/3. Estimated by the Kaplan-Meier method and a 2-sided 95% CI for median was computed using the Brookmeyer and Crowley method.
Time Frame: Days 8, 15, 22, 29, 36, 43; Weeks 7, 13, 25, 37; at Week 4, 19, 31 (only stratum 2/3); then every 12 weeks upto 24 months; then once/year; until criteria was first met for CHR (maximum participant time to first CHR of 65 days).
Population: All treated participants with CHR in strata 1 and 2/3.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose: Participants with imatinib-resistant Philadelphia chromosome positive (Ph+) chronic myeloid leukemia (CML) in chronic phase (CP). Starting Dose Level of 60 mg/m^2; Escalated/Dose level 2 of 80 mg/m^2 QD, as long as clinical benefit was maintained.
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose
Number analyzed (Participants) | 16 | 6
days | 21.5 [16.0 to 23.0] | 39.5 [36.0 to 44.0]

21. Secondary Outcome: Duration of Major Hematologic Response (MaHR): Stratum 2/3 (Ph+ALL or AP/BP-CML)
Description: Duration of MaHR is the time (in months) from the first day criteria were met for MaHR, provided they were confirmed later at least after 28 days with no concomitant use of anagrelide or hydroxyurea during this interval, until death or progression was first observed. MaHR: Defined as participants having as best response a CHR or CHRp. Refer to outcome measure 20 for criteria for CHR or CHRp. The Kaplan-Meier plot was used. A 2-sided, 95% CI for the median was computed using the Brookmeyer and Crowley method.
Time Frame: From the date of first confirmed MaHR to date of progression, death, or last tumor assessment (maximum participant duration of response of 37 months).
Population: All treated participants with MaHR in stratum 2/3. Participants who neither discontinued due to progression nor progressed nor died were censored on the date of their last hematologic or cytogenetic assessment, whichever came last.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose
Number analyzed (Participants) | 8
months | 4.4 [3.5 to NA] — Upper limit could not be derived with the method of Brookmeyer and Crowley.

22. Secondary Outcome: Duration of Complete Hematologic Response (CHR): Stratum 1 (Ph+ CP-CML) and Stratum 2/3 (Ph+ALL or AP/BP-CML)
Description: Duration of CHR is the time (in months) from the first day criteria were met for CHR, provided they were confirmed later (after 28 days) with no concomitant use of anagrelide or hydroxyurea during this interval until death or progression was first observed. Refer to Outcome Measure 20 for criteria for CHR (Stratum 1) and Outcome Measure 19 for CHR (Stratum 2/3). The Kaplan-Meier plot was used. A 2-sided, 95% CI for the median was computed using the Brookmeyer and Crowley method.
Time Frame: From the date of first confirmed CHR to date of progression, death, or last tumor assessment (maximum participant duration of response of 50 months).
Population: Treated participants with CHR in strata 1 and 2/3. Participants who neither discontinued due to progression nor progressed nor died were censored on the date of their last hematologic or cytogenetic assessment, whichever came last.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose
Number analyzed (Participants) | 16 | 6
months | NA [14.3 to NA] — Median duration of CHR was not estimable as only 5 participants had disease progression and more than 50% of participants were censored. | 7.3 [3.5 to NA] — Upper limit could not be derived with the method of Brookmeyer and Crowley.

23. Secondary Outcome: Percentage of Participants With Confirmed Hematologic Response (HR) at Recommended Phase II Dose: Stratum 1 (Ph+ CP-CML)
Description: A participant was said to have a confirmed HR if all the criteria for HR were fulfilled again at least 28 days after they first met with no concomitant use of anagrelide or hydroxyurea during this interval. HR observed in stratum 1 was CHR. Refer to Outcome Measure 20 for criteria for CHR. The Clopper and Pearson method was used to compute 95% exact CIs.
Time Frame: as for outcome 16
Population: All treated participants in stratum 1 who received at least 1 dose of dasatinib 60 mg/m^2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Stratum1 Ph+ CP-CML (Dasatinib 60 mg/m^2): Participants with imatinib-resistant Philadelphia chromosome positive (Ph+) chronic myeloid leukemia (CML) in chronic phase (CP). Dasatinib 60 mg/m^2 QD, as long as clinical benefit was maintained.
Arm/Group | Stratum1 Ph+ CP-CML (Dasatinib 60 mg/m^2)
Number analyzed (Participants) | 11
percentage of participants | 90.9 [58.7 to 99.8]

24. Secondary Outcome: Percentage of Participants With Confirmed Hematologic Response (HR) at Recommended Phase II Dose: Stratum 2/3 (Ph+ALL or AP/BP-CML)
Description: A participant is said to have a confirmed HR if criteria for HR were fulfilled again at least 28 days after they first met with no concomitant use of anagrelide or hydroxyurea during this interval. Confirmed HR observed in stratum 2/3 was either CHR or MaHR or overall hematologic response (OHR). Refer to Outcome Measure 19 for criteria for CHR and MaHR. OHR is defined as MaHR or MiHR. MiHR=CHRp except blasts in BM (≥ 5% and ≤ 15% blasts in BM). The Clopper and Pearson method was used to compute 95% exact CIs.
Time Frame: Days 8, 15, 22, 29, 36, 43; Weeks 4, 7, 13, 19, 25, 31, 37; then every 12 weeks upto 24 months; then once/year; EOT (Median duration of therapy in months: Stratum 2/3=3.02 [Range: 0.53-37.72])
Population: All treated participants in stratum 2/3: Participants who received at least 1 dose of dasatinib 80 mg/m^2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 80 mg/m^2)
Number analyzed (Participants) | 9
percentage of participants
  CHR | 55.6 [21.2 to 86.3]
  MaHR | 66.7 [29.9 to 92.5]
  OHR | 66.7 [29.9 to 92.5]

25. Secondary Outcome: Number of Participants With Molecular Responses in Stratum 1 (Ph+ CP-CML)
Description: Molecular response was calculated by measuring p210 variant of BCR-ABL transcripts in blood during treatment using quantitative polymerase chain reaction (qPCR) assay. Major molecular response (MMR): Ratio of the BCR-ABL to ABL <10^-3 or 0.1% on the international scale. Complete molecular response (CMR): Complete absence of BCR-ABL or the ratio is <10^-4.5 or 0.00316% on the international scale. Confirmed MMR or CMR = Criteria met again >6 weeks. BCR-ABL=the fused gene found in participants with this type of CML.
Time Frame: At baseline (within 3 weeks before initiation of study therapy), After hematologic response, EOT (Median duration of therapy in months: Stratum 1=24.11 [Range: 2.27-50.63])
Population: All treated participants in stratum 1: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum 1 Ph+ CP-CML (Dasatinib 60 mg/m^2) | Stratum 1 Ph+ CP-CML (Dasatinib 80 mg/m^2)
Number analyzed (Participants) | 11 | 6
participants
  MMR (Overall) | 6 | 2
  CMR (Unconfirmed) | 3 | 1
  CMR (Confirmed) | 1 | 0

26. Secondary Outcome: Number of Participants With Major Molecular Response (MMR) in Stratum 2/3 (Ph+ ALL or AP/BP-CML)
Description: Molecular response was calculated by measuring BCR-ABL transcripts in blood during treatment using qPCR assay. MMR: Ratio of the BCR-ABL to ABL <10^-3 or a ≥3 log reduction from baseline in participants with p190 variant; ratio of the BCR-ABL to ABL <10^-3 on the international scale in participants with p210 variant. BCR-ABL=the fused gene found in participants with this type of CML.
Time Frame: At baseline (within 3 weeks before initiation of study therapy), After hematologic response, EOT (Median duration of therapy in months: Stratum 2/3=3.02 [Range: 0.53-37.72])
Population: All treated participants (14 with p190 variant and 3 with p210 variant BCR-ABL transcripts) in stratum 2/3: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 60 mg/m^2) | Stratum 2/3 Ph+ ALL or AP/BP-CML (Dasatinib 80 mg/m^2)
Number analyzed (Participants) | 8 | 9
participants | 2 | 6

27. Secondary Outcome: Progression Free Survival (PFS)
Description: Time in months from 1st first dose until progression (resistance or refractory disease) or death was first documented by investigator. Progressive disease: Resistant disease for which investigator may electively stop treatment or refractory disease requiring cessation of study treatment. The PFS was estimated using the Kaplan-Meier product-limit method, and a two-sided 95% CI for the median PFS time was computed using the method of Brookmeyer and Crowley.
Time Frame: From the date of randomization to date of progression, death, last tumor assessment, or 5 years after EOT (Median duration of therapy in months: Stratum 1=24.11 [Range: 2.27-50.63]; Stratum 2/3=3.02 [Range: 0.53-37.72]; Stratum 4=1.14 [Range: 0.03-3.38])
Population: All treated participants: Participants who received at least 1 dose of study therapy. If no progression or death was reported, PFS was censored at the last assessment date done on-study (i.e., up to 30 days after last dosing date) at which non-progression was reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose | Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose
Number analyzed (Participants) | 17 | 17 | 24
months | 53.6 [11.4 to NA] — Upper limit not reached | 4.9 [0.6 to 8.4] | 1.4 [0.4 to 1.6]

28. Secondary Outcome: Overall Survival (OS)
Description: Defined as time in months from start of study therapy to death. The OS was estimated using the Kaplan-Meier product-limit method, and a two-sided 95% CI for the median OS time was computed using the Brookmeyer and Crowley method.
Time Frame: From start of study therapy until death or 5 years after EOT (Median duration of therapy in months: Stratum 1=24.11 [Range: 2.27-50.63]; Stratum 2/3=3.02 [Range: 0.53-37.72]; Stratum 4=1.14 [Range: 0.03-3.38])
Population: All treated participants: Participants who received at least 1 dose of study therapy. Participants lost to followup were censored on the last date the participant was known to be alive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose | Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose
Number analyzed (Participants) | 17 | 17 | 24
months | NA [NA to NA] — Median OS was not estimable as 14 of the 17 participants were censored by 25 May 2011 | 8.6 [3.2 to NA] — Upper limit not reached | 3.0 [1.7 to 4.4]

29. Secondary Outcome: Dasatinib Plasma Pharmacokinetic (PK) Parameter: Time to Achieve the Observed Maximum Plasma Concentration (Tmax) by Age Group
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. Tmax is the time taken to reach the maximum observed plasma concentration.
Time Frame: During Week 1 of Course 1, and any course in which dose escalation was performed (at pre-dose, and at 0.5, 1, 2, 4, 6, 8 and 24 hours).
Population: All treated participants with plasma samples available. Each participant could have 1, 2, or 3 plasma PK profiles sampled, depending on the number of times the dose of dasatinib was escalated. n=number of PK parameters included.
Measure: Median (Full Range); unit: hours
Groups:
- Dasatinib 60 mg/m^2 QD Starting Dose: Stratum 1 (Ph+ CP-CML): Participants with imatinib-resistant Ph+ CML in CP; Stratum 2/3 (PH+ ALL OR AP/BP-CML): Participants with imatinib-resistant or imatinib-intolerant Ph+ CML in AP, or in MBP, or in LBP; or relapsed or refractory Ph+ ALL after imatinib use; or second or subsequent relapse of Ph+ AML; Stratum 4 (PH- ALL/AML): Participants with second or subsequent relapse of Ph- ALL or Ph- AML. Strata 1, 2/3, and 4: 60 mg/m^2 starting dose; 80 mg/m^2 escalated/dose level 2; Stratum 4: 100 mg/m^2 escalated/dose level 3 and 120 mg/m^2 escalated/dose level 4. QD, as long as clinical benefit was observed.
Arm/Group | Dasatinib 60 mg/m^2 QD Starting Dose
Number analyzed (Participants) | 53
hours
  Infants and Toddlers (age<2 years old; n=2) | 0.5 (0.0) [0.5 to 0.5]
  Children (age>=2 and <12 years old; n=43) | 1.1 (58.6) [0.5 to 4.1]
  Adolescents (age>=12 and <18 years old; n=28) | 1.0 (82.2) [0.5 to 6.0]
  Above 18 Years (n=1) | 0.9 (NA) [0.9 to 0.9]
  Total (n=74) | 1.0 (70.9) [0.5 to 6.0]

30. Secondary Outcome: Dasatinib Plasma Pharmacokinetic Parameter: Terminal Half-life (T 1/2) by Age Group
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. T 1/2 is the time required for the concentration of the drug to reach half of its original value in plasma.
Time Frame: as for outcome 29
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Groups:
- Dasatinib 60 mg/m^2 QD Starting Dose: Stratum 1 (Ph+ CP-CML): Participants with imatinib-resistant Ph+ CML in CP; Stratum 2/3 (PH+ ALL OR AP/BP-CML): Participants with imatinib-resistant or imatinib-intolerant Ph+ CML in AP, or in MBP, or in LBP; or relapsed or refractory Ph+ ALL after imatinib use; or second or subsequent relapse of Ph+ AML; Stratum 4 (PH- ALL/AML): Participants with second or subsequent relapse of Ph- ALL or Ph- AML. Tablets, Oral; If necessary in participants who could not swallow, tablets were dispersed into 30 cc of 100% fruit juice with no preservatives (minute maid lemonade or orange juice or apple juice). Strata 1, 2/3, and 4: 60 mg/m^2 starting dose; 80 mg/m^2 escalated/dose level 2; Stratum 4: 100 mg/m^2 escalated/dose level 3 and 120 mg/m^2 escalated/dose level 4. QD, as long as clinical benefit was observed.
Arm/Group | Dasatinib 60 mg/m^2 QD Starting Dose
Number analyzed (Participants) | 53
hours
  Infants and Toddlers (age<2 years old; n=2) | 2.1 (24.0)
  Children (age>=2 and <12 years old; n=36) | 3.0 (62.8)
  Adolescents (age>=12 and <18 years old; n=22) | 3.8 (43.9)
  Above 18 years (n=1) | 7.3 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated.
  Total (n=61) | 3.3 (55.7)

31. Secondary Outcome: Dasatinib Plasma Pharmacokinetic Parameter: Dose Normalized Observed Maximum Plasma Concentration (Cmax) by Age Group
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. Dose Normalized Cmax is the maximum observed concentration of drug substance in plasma normalized for different dasatinib dose levels.
Time Frame: as for outcome 29
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg/m^2
Arm/Group | Dasatinib 60 mg/m^2 QD Starting Dose
Number analyzed (Participants) | 53
ng/mL/mg/m^2
  Infants and Toddlers (age<2 years old; n=2) | 1.0 (15.2)
  Children (age>=2 and <12 years old; n=43) | 1.9 (79.9)
  Adolescents (age>=12 and <18 years old; n=28) | 1.0 (69.7)
  Above 18 Years (n=1) | 0.9 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated.
  Total (n=74) | 1.5 (86.9)

32. Secondary Outcome: Dasatinib Plasma Pharmacokinetic Parameter: Dose Normalized Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC[0-T]) by Age Group
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. AUC[0-T] is the area under the plasma concentration-time curve from time zero to time of last quantifiable concentration, normalized by dasatinib dose level.
Time Frame: as for outcome 29
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL/mg/m^2
Arm/Group | Dasatinib 60 mg/m^2 QD Starting Dose
Number analyzed (Participants) | 53
ng.h/mL/mg/m^2
  Infants and Toddlers (age<2 years old; n=2) | 2.8 (4.6)
  Children (age>=2 and <12 years old; n=40) | 6.1 (95.7)
  Adolescents (age>=12 and <18 years old; n=28) | 3.8 (66.8)
  Above 18 Years (n=1) | 2.2 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated.
  Total (n=71) | 4.9 (98.1)

33. Secondary Outcome: Dasatinib Plasma Pharmacokinetic Parameter: Dose Normalized Area Under the Plasma Concentration Versus Time Curve From Time Zero Extrapolated to Infinite Time (AUC[INF]) by Age Group
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. AUC (0-inf) is the area under the plasma concentration-time curve from time zero extrapolated to infinite time, normalized by dasatinib dose level.
Time Frame: as for outcome 29
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL/mg/m^2
Arm/Group | Dasatinib 60 mg/m^2 QD Starting Dose
Number analyzed (Participants) | 53
ng.h/mL/mg/m^2
  Infants and Toddlers (age<2 years old; n=2) | 3.2 (17.7)
  Children (age>=2 and <12 years old; n=36) | 6.7 (95.0)
  Adolescents (age>=12 and <18 years old; n=22) | 4.2 (67.6)
  Above 18 Years (n=1) | 2.4 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated.
  Total (n=61) | 5.4 (97.1)

34. Secondary Outcome: Dasatinib Plasma Pharmacokinetic Parameter: Observed Maximum Plasma Concentration (Cmax) by Dose Level and Age Group
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. Cmax is the maximum observed concentration of drug substance in plasma.
Time Frame: as for outcome 29
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Dasatinib 60 mg/m^2: Dasatinib 60 mg/m^2 QD, as long as clinical benefit was maintained.
- Dasatinib 80 mg/m^2: Tablets, Oral; If necessary in participants who could not swallow, tablets were dispersed into 30 cc of 100% fruit juice with no preservatives (minute maid lemonade or orange juice or apple juice). Dasatinib 80 mg/m^2 QD, as long as clinical benefit was maintained.
- Dasatinib 100 mg/m^2: Tablets, Oral; If necessary in participants who could not swallow, tablets were dispersed into 30 cc of 100% fruit juice with no preservatives (minute maid lemonade or orange juice or apple juice). Dasatinib 100 mg/m^2 QD, as long as clinical benefit was maintained.
- Dasatinib 120 mg/m^2: Tablets, Oral; If necessary in participants who could not swallow, tablets were dispersed into 30 cc of 100% fruit juice with no preservatives (minute maid lemonade or orange juice or apple juice). Dasatinib 120 mg/m^2 QD, as long as clinical benefit was maintained.
Arm/Group | Dasatinib 60 mg/m^2 | Dasatinib 80 mg/m^2 | Dasatinib 100 mg/m^2 | Dasatinib 120 mg/m^2
Number analyzed (Participants) | 20 | 25 | 19 | 10
ng/mL
  Infants and Toddlers (age>2yr; n=0; n=0; n=1; n=1) | NA (NA) — No participants in this age group. | NA (NA) — No participants in this age group. | 30.6 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated. | 53.8 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated.
  Children (age>=2 & <12yr; n=11; n=16; n=9; n=7) | 110.6 (61.8) | 142.5 (80.2) | 111.2 (82.6) | 208.4 (78.5)
  Adolescents (age>=12; n=9; n=8; n=9; n=2) | 92.6 (50.6) | 116.5 (73.0) | 235.1 (59.0) | 123.3 (68.3)
  Above 18 years (n=0; n=1; n=0; n=0) | NA (NA) — No participants in this age group. | 143.2 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated. | NA (NA) — No participants in this age group. | NA (NA) — No participants in this age group.
  Total | 102.1 (58.0) | 133.6 (77.6) | 148.1 (75.0) | 163.9 (87.6)

35. Secondary Outcome: Dasatinib Plasma Pharmacokinetic (PK) Parameter: Time to Achieve the Observed Maximum Plasma Concentration (Tmax) By Dose Level and Age Group
Description: as for outcome 29
Time Frame: as for outcome 29
Population: All treated participants with plasma samples available. Each participant could have more than 1 plasma profiles sampled, depending on the number of times the dose of dasatinib was escalated. n=number of PK parameters included.
Measure: Median (Full Range); unit: hour
Arm/Group | Dasatinib 60 mg/m^2 | Dasatinib 80 mg/m^2 | Dasatinib 100 mg/m^2 | Dasatinib 120 mg/m^2
Number analyzed (Participants) | 20 | 25 | 19 | 10
hour
  Infants and Toddlers (age<2yr; n=0; n=0; n=1; n=1) | NA (NA) [NA to NA] — No participants in this age group. | NA [NA to NA] — No participants in this age group. | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 0.5]
  Children (age>=2 & <12yr; n=11; n=16; n=9; n=7) | 1.1 (61.8) [0.5 to 2.1] | 1.5 [0.5 to 3.2] | 1.1 [0.6 to 4.1] | 1.0 [0.9 to 2.2]
  Adolescents (age>=12 & <12yr; n=9; n=8; n=9; n=2) | 1.0 [0.5 to 4.0] | 1.1 [0.5 to 4.0] | 1.0 [0.5 to 6.0] | 1.6 [1.0 to 2.1]
  Above 18 years (n=0; n=1; n=0; n=0) | NA [NA to NA] — No participants in this age group. | 0.9 [0.9 to 0.9] | NA [NA to NA] — No participants in this age group. | NA [NA to NA] — No participants in this age group.
  Total | 1.0 [0.5 to 4.0] | 1.1 [0.5 to 4.0] | 1.0 [0.5 to 6.0] | 1.0 [0.5 to 2.2]

36. Secondary Outcome: Dasatinib Plasma Pharmacokinetic Parameter: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC[0-T]) by Dose Level and Age Group
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. AUC(0-T) is the area under the plasma concentration-time curve from time zero to time of last quantifiable concentration.
Time Frame: as for outcome 29
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Dasatinib 60 mg/m^2 | Dasatinib 80 mg/m^2 | Dasatinib 100 mg/m^2 | Dasatinib 120 mg/m^2
Number analyzed (Participants) | 19 | 25 | 18 | 9
ng.h/mL
  Infants and Toddlers (age<2yr; n=0; n=0; n=1; n=1) | NA (NA) [NA to NA] — No participants in this age group. | NA (NA) — No participants in this age group. | 100.8 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated. | 134.9 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated.
  Children (age>=2 & <12yr; n=10; n=16; n=8; n=6) | 295.0 (63.5) | 490.8 (96.7) | 373.5 (82.0) | 676.7 (99.9)
  Adolescents (age>=12 & <18yr; n=9; n=8; n=9; n=2) | 320.8 (59.1) | 488.1 (35.0) | 787.0 (76.2) | 526.1 (56.6)
  Above 18 years (n=0; n=1; n=0; n=0) | NA (NA) — No participants in this age group. | 367.2 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated. | NA (NA) — No participants in this age group. | NA (NA) — No participants in this age group.
  Total | 307.0 (60.2) | 484.3 (88.9) | 504.1 (89.6) | 534.9 (103.9)

37. Secondary Outcome: Dasatinib Plasma Pharmacokinetic Parameter: Area Under the Plasma Concentration Versus Time Curve From Time Zero Extrapolated to Infinite Time (AUC[INF]) by Dose Level and Age Group
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. AUC(INF) is the area under the plasma concentration-time curve from time zero extrapolated to infinite time.
Time Frame: as for outcome 29
Population: All treated participants with plasma samples available. n=number of PK parameters included. Each participant could have more than 1 plasma profiles sampled, depending on the number of times the dose of dasatinib was escalated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Dasatinib 60 mg/m^2 | Dasatinib 80 mg/m^2 | Dasatinib 100 mg/m^2 | Dasatinib 120 mg/m^2
Number analyzed (Participants) | 18 | 20 | 15 | 8
ng.h/mL
  Infants and Toddlers (age<2yr; n=0; n=0; n=1; n=1) | 0 (0) | 0 (0) | 127.7 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated. | 142.1 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated.
  Children (age>=2 & <12yr; n=10; n=14; n=7; n=5) | 313.9 (59.8) | 513.6 (99.2) | 429.1 (76.8) | 817.6 (93.7)
  Adolescents (age>=12 & <18yr; n=8; n=5; n=7; n=2) | 305.8 (60.9) | 605.1 (25.3) | 1008.9 (69.4) | 547.8 (58.2)
  Above 18 years (n=0; n=1; n=0; n=0) | 0 (0) | 390.0 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated. | 0 (0) | 0 (0)
  Total | 310.3 (58.6) | 527.8 (90.4) | 589.8 (86.2) | 594.4 (101.5)

38. Secondary Outcome: Dasatinib Plasma Pharmacokinetic Parameter: Terminal Half-life (T 1/2) by Dose Level and Age Group
Description: as for outcome 30
Time Frame: as for outcome 29
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Dasatinib 60 mg/m^2 | Dasatinib 80 mg/m^2 | Dasatinib 100 mg/m^2 | Dasatinib 120 mg/m^2
Number analyzed (Participants) | 18 | 20 | 15 | 8
hour
  Infants and Toddlers (age<2yr; n=0; n=0; n=1; n=1) | NA (NA) — No participants in this age group. | NA (NA) — No participants in this age group. | 2.5 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated. | 1.8 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated.
  Children (age>=2 & <12yr; n=10; n=14; n=7; n=5) | 2.4 (1.0) | 3.9 (1.9) | 4.6 (3.5) | 3.2 (1.9)
  Adolescents (age>=12 & <18yr; n=8; n=5; n=7; n=2) | 3.7 (1.6) | 5.1 (0.5) | 4.5 (2.5) | 3.5 (2.9)
  Above 18 years (n=0; n=1; n=0; n=0) | NA (NA) — No participants in this age group. | 7.3 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated. | NA (NA) — No participants in this age group. | NA (NA) — No participants in this age group.
  Total | 3.0 (1.4) | 4.4 (1.8) | 4.4 (2.9) | 3.1 (1.9)

39. Secondary Outcome: Dasatinib Metabolite (BMS-582691) Plasma Pharmacokinetic Parameter: Observed Maximum Plasma Concentration (Cmax) by Dose Level and Age Group
Description: as for outcome 34
Time Frame: as for outcome 29
Population: All treated participants with plasma samples available. n=number of PK parameters included. Each participant could have 1, 2, or 3 plasma PK profiles sampled, depending on the number of times the dose of dasatinib was escalated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dasatinib 60 mg/m^2 | Dasatinib 80 mg/m^2 | Dasatinib 100 mg/m^2 | Dasatinib 120 mg/m^2
Number analyzed (Participants) | 18 | 25 | 16 | 10
ng/mL
  Infants and Toddlers (age<2yr; n=0; n=0; n=0; n=1) | NA (NA) — No participants in this age group. | NA (NA) — No participants in this age group. | NA (NA) — No participants in this age group. | 1.2 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated.
  Children (age>=2 & <12yr; n=10; n=16; n=7; n=7) | 3.6 (46.4) | 3.4 (82.0) | 6.0 (69.3) | 4.8 (65.3)
  Adolescents (age>=12 & <18yr; n=8; n=8; n=9; n=2) | 3.1 (40.3) | 3.6 (56.7) | 6.9 (75.0) | 4.3 (77.9)
  Above 18 years (n=0; n=1; n=0; n=0) | NA (NA) — No participants in this age group. | 2.2 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated. | NA (NA) — No participants in this age group. | NA (NA) — No participants in this age group.
  Total | 3.4 (43.7) | 3.4 (74.4) | 6.5 (72.0) | 4.1 (70.8)

40. Secondary Outcome: Dasatinib Metabolite (BMS-582691) Plasma Pharmacokinetic (PK) Parameter: Time to Achieve the Observed Maximum Plasma Concentration (Tmax) By Dose Level and Age Group
Description: as for outcome 29
Time Frame: as for outcome 29
Population: as for outcome 37
Measure: Median (Full Range); unit: hour
Arm/Group | Dasatinib 60 mg/m^2 | Dasatinib 80 mg/m^2 | Dasatinib 100 mg/m^2 | Dasatinib 120 mg/m^2
Number analyzed (Participants) | 18 | 25 | 16 | 10
hour
  Infants and Toddlers (age<2yr; n=0; n=0; n=0; n=1) | NA [NA to NA] — No participants in this age group. | NA [NA to NA] — No participants in this age group. | NA [NA to NA] — No participants in this age group. | 0.9 [0.9 to 0.9]
  Children (age>=2 & <12yr; n=10; n=16; n=7; n=7) | 2.0 [1.0 to 4.5] | 2.0 [0.5 to 6.0] | 2.1 [1.0 to 4.1] | 2.0 [1.0 to 2.2]
  Adolescents (age>=12 & <18yr ; n=8; n=8; n=9; n=2) | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 8.1] | 2.1 [2.0 to 2.1]
  Above 18 years (n=0; n=1; n=0; n=0) | NA [NA to NA] — No participants in this age group. | 0.9 [0.9 to 0.9] | NA [NA to NA] — No participants in this age group. | NA [NA to NA] — No participants in this age group.
  Total | 2.0 [1.0 to 4.5] | 2.0 [0.5 to 6.0] | 2.0 [1.0 to 8.1] | 2.0 [0.9 to 2.2]

41. Secondary Outcome: Dasatinib Metabolite (BMS-582691) Plasma Pharmacokinetic Parameter: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC[0-T]) by Dose Level and Age Group
Description: as for outcome 36
Time Frame: as for outcome 29
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Dasatinib 60 mg/m^2 | Dasatinib 80 mg/m^2 | Dasatinib 100 mg/m^2 | Dasatinib 120 mg/m^2
Number analyzed (Participants) | 13 | 21 | 14 | 9
ng.h/mL
  Infants and Toddlers (age<2yr; n=0; n=0; n=0; n=1) | NA (NA) — No participants in this age group. | NA (NA) — No participants in this age group. | NA (NA) — No participants in this age group. | 1.9 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated.
  Children (age>=2 & <12yr; n=7; n=12; n=5; n=6) | 8.8 (50.4) | 16.6 (145.2) | 25.4 (71.1) | 23.6 (102.2)
  Adolescents (age>=12 & <12yr; n=6; n=8; n=9; n=2) | 12.3 (38.4) | 13.5 (54.4) | 20.0 (112.3) | 15.8 (105.5)
  Above 18 years (n=0; n=1; n=0; n=0) | NA (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated. | 6.6 (NA) — Due to insufficient number of participants in this age group (only 1 participant), CV% could not be calculated. | NA (NA) — No participants in this age group. | NA (NA) — No participants in this age group.
  Total | 10.3 (44.9) | 14.7 (141.1) | 21.8 (100.1) | 16.3 (110.3)

42. Secondary Outcome: Concentration of Dasatinib in Cerebrospinal Fluid (CSF) by Dose Level and Age Group
Description: Concentration of dasatinib in CSF was assessed only in participants who had lumbar puncture during the treatment. y=years
Time Frame: 4 hours after oral dose
Population: All treated participants with CSF samples available. n=number of PK parameters included. Each participant could have more than 1 CSF profiles sampled, depending on the number of times the dose of dasatinib was escalated.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dasatinib 60 mg/m^2 | Dasatinib 80 mg/m^2 | Dasatinib 100 mg/m^2 | Dasatinib 120 mg/m^2
Number analyzed (Participants) | 4 | 10 | 6 | 1
ng/mL
  Children (age>=2 & <12 y; n=3, n=9, n=3, n=1) | 1.1 (0.2) | 1.5 (0.6) | 1.7 (0.4) | 3.8 (NA) — Due to insufficient number of participants in this age group (only 1 participant), standard deviation could not be calculated.
  Adolescents (age>=12 & <18 y; n=1; n=1; n=3; n=0) | 1.1 (NA) — Due to insufficient number of participants in this age group (only 1 participant), standard deviation could not be calculated. | 1.0 (NA) — Due to insufficient number of participants in this age group (only 1 participant), standard deviation could not be calculated. | 2.6 (0.6) | NA (NA) — No participants in this age group.
  Total (Children + Adolescents;n=4; n=10; n=6; n=1) | 1.1 (0.1) | 1.4 (0.6) | 2.1 (0.7) | 3.8 (NA) — Due to insufficient number of participants in this age group (only 1 participant), standard deviation could not be calculated.

43. Secondary Outcome: Number of Participants With BCR-ABL Mutations at Baseline: Stratum1 Ph+ CP-CML and Stratum 2/3 Ph+ALL or AP/BP-CML
Description: BCR-ABL, also referred to as the Philadelphia chromosome, is formed from the fusion of the BCR gene on chromosome 22 with the ABL gene on chromosome 9.
Time Frame: At baseline (within 3 weeks before initiation of study therapy)
Population: All treated participants in strata 1 and 2/3: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose
Number analyzed (Participants) | 17 | 17
participants
  L384M | 1 | 0
  G250E | 1 | 0
  T315I | 0 | 1
  Y253H | 0 | 1
  Y253F | 0 | 1
  No Mutation | 15 | 11
  No Data | 0 | 3

44. Other Pre Specified Outcome: Number of Participants With Hematologic Toxicity at Baseline by NCI CTCAE Version 3.0
Description: GR1=Mild; GR2=Moderate; GR3=Severe; GR4=Life-threatening or disabling. Normal ranges provided by local laboratory and may also vary from site to site. White Blood Cell (WBC):GR1=<LLN-3.0*10^9/L; GR2=<3.0-2.0*10^9/L; GR3=<2.0-1.0*10^9/L; GR4=<1.0*10^9/L. Absolute Neutrophil Count (ANC): GR1=<LLN-1.5*10^9 /L; GR2=<1.5-1.0*10^9/L; GR3=<1.0-0.5*10^9/L; GR4=<0.5*10^9/L. Hemoglobin: GR1=<LLN-10.0g/dL; GR2=<10.0-8.0g/dL; GR3=<8.0-6.5g/dL; GR4=<6.5g/dL. Platelets: GR1=<LLN-75.0*10^9/L; GR2=<75.0-50.0*10^9/L; GR3=<50.0-25.0*10^9/L; GR4=<25.0*10^9/L. LLN=lower limit of normal.
Time Frame: At baseline (within 1 week before initiation of study therapy)
Population: All treated participants: Participants who received at least one dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose | Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose
Number analyzed (Participants) | 17 | 17 | 24
participants
  WBC GR1 | 1 | 2 | 3
  WBC GR2 | 0 | 2 | 2
  WBC GR3 | 0 | 0 | 6
  WBC GR4 | 0 | 1 | 4
  ANC GR1 | 1 | 2 | 3
  ANC GR2 | 1 | 1 | 0
  ANC GR3 | 0 | 2 | 3
  ANC GR4 | 0 | 2 | 13
  Platelet GR1 | 1 | 5 | 5
  Platelet GR2 | 0 | 2 | 3
  Platelet GR3 | 0 | 3 | 8
  Platelet GR4 | 0 | 2 | 6
  Hemoglobin GR1 | 7 | 7 | 7
  Hemoglobin GR2 | 1 | 7 | 7
  Hemoglobin GR3 | 0 | 1 | 3
  Hemoglobin GR4 | 0 | 0 | 0

45. Other Pre Specified Outcome: Number of Participants With Serum Chemistry Abnormalities (Liver and Renal Function) at Baseline by NCI CTCAE Version 3.0
Description: GR1=Mild; GR2=Moderate; GR3=Severe; GR4=Life-threatening or disabling. Normal ranges provided by local laboratory and may also vary from site to site. Aspartate aminotransferase (AST) and alanine aminotransferase(ALT): GR1=>ULN-2.5*ULN; GR2=>2.5-5.0*ULN; GR3=>5.0-20.0*ULN; GR4=>20.0*ULN. Total bilirubin:GR1=>ULN-1.5*ULN, GR2=>1.5-3.0*ULN, GR3=>3-10*ULN, GR4=>10*ULN. Creatinine: GR1=>ULN-1.5*ULN, GR2=>1.5-3.0*ULN, GR3=>3.0-6.0*ULN, GR4=>6.0*ULN. ULN=upper limit of normal.
Time Frame: At baseline (within 1 week before initiation of study therapy)
Population: All treated participants: Participants who received at least one dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose | Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose
Number analyzed (Participants) | 17 | 17 | 24
participants
  AST GR1 | 1 | 3 | 8
  AST GR2 | 0 | 2 | 1
  AST GR3 | 0 | 1 | 0
  AST GR4 | 0 | 0 | 0
  AST GR Not Reported | 1 | 3 | 2
  High ALT GR1 | 2 | 6 | 6
  High ALT GR2 | 0 | 2 | 5
  High ALT GR3 | 0 | 0 | 0
  High ALT GR4 | 0 | 0 | 0
  High ALT GR Not Reported | 0 | 0 | 0
  High Total Bilirubin GR1 | 3 | 0 | 1
  High Total Bilirubin GR2 | 0 | 1 | 0
  High Total Bilirubin GR3 | 0 | 0 | 0
  High Total Bilirubin G4 | 0 | 0 | 0
  High Total Bilirubin GR Not Reported | 0 | 0 | 1
  High Serum Creatinine GR1 | 2 | 0 | 4
  High Serum Creatinine GR2 | 0 | 1 | 0
  High Serum Creatinine GR3 | 0 | 0 | 0
  High Serum Creatinine GR4 | 0 | 0 | 0
  High Serum Creatinine GR Not Reported | 0 | 0 | 1

46. Other Pre Specified Outcome: Number of Participants With Serum Chemistry Abnormalities (Calcium, Magnesium, and Phosphate) at Baseline by NCI CTCAE Version 3.0
Description: as for outcome 5
Time Frame: At baseline (within 1 week before initiation of study therapy)
Population: All treated participants: Participants who received at least one dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose | Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose
Number analyzed (Participants) | 17 | 17 | 24
participants
  Low Calcium GR1 | 0 | 0 | 1
  Low Calcium GR2 | 0 | 0 | 0
  Low Calcium GR3 | 0 | 0 | 0
  Low Calcium GR4 | 0 | 0 | 0
  Low Calcium GR Not Reported | 0 | 0 | 2
  Low Magnesium GR1 | 0 | 6 | 0
  Low Magnesium GR2 | 0 | 0 | 0
  Low Magnesium GR3 | 0 | 0 | 0
  Low Magnesium GR4 | 0 | 0 | 0
  Low Magnesium GR Not Reported | 0 | 0 | 2
  Low Phosphate GR1 | 0 | 1 | 0
  Low Phosphate GR2 | 0 | 0 | 0
  Low Phosphate GR3 | 0 | 1 | 0
  Low Phosphate GR4 | 0 | 0 | 0
  Low Phosphate GR Not Reported | 2 | 0 | 2

47. Secondary Outcome: Number of Participants With BCR-ABL Mutations at End-of-Treatment: Stratum1 Ph+ CP-CML and Stratum2/3 Ph+ ALL or AP/BP-CML
Description: BCR-ABL = These are fused genes found in participants with this type of leukemia.
Time Frame: At EOT (Median duration of therapy in months: Stratum 1=24.11 [Range: 2.27-50.63]; Stratum 2/3=3.02 [Range: 0.53-37.72])
Population: All treated participants in strata 1 and 2/3: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose
Number analyzed (Participants) | 17 | 17
participants
  T315I | 0 | 4
  No Mutation | 8 | 9
  No Data | 9 | 4

48. Secondary Outcome: Number of Participants With FLT3 and KIT Mutations in Stratum4 Ph- ALL/AML at Baseline
Description: FLT3 and KIT = These are fused genes found in participants with this type of leukemia.
Time Frame: At baseline (within 3 weeks before initiation of study therapy)
Population: All treated participants in stratum 4: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose
Number analyzed (Participants) | 24
participants
  FLT3 Absent | 20
  FLT3 Present | 1
  FLT3 No Data | 3
  KIT Absent | 21
  KIT Present | 0
  KIT No Data | 3

49. Secondary Outcome: Number of Participants With FLT3 and KIT Mutations in Stratum4 Ph- ALL/AML at End-Of-Treatment
Description: FLT3 and KIT = These are fused genes found in participants with this type of leukemia.
Time Frame: At EOT (Median duration of therapy in months: Stratum 4=1.14 [Range: 0.03-3.38])
Population: All treated participants in stratum 4: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose
Number analyzed (Participants) | 24
participants
  FLT3 Absent | 6
  FLT3 Present | 0
  FLT3 No Data | 18
  KIT Absent | 6
  KIT Present | 0
  KIT No Data | 18

ADVERSE EVENTS:
Time Frame: From first dose to 100 days post last dose
Arm/Group | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose | Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose
Serious Adverse Events (participants affected / at risk) | 8/17 | 14/17 | 22/24
Other Adverse Events (participants affected / at risk) | 16/17 | 16/17 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose (N=17) | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose (N=17) | Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose (N=24)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Performance status decreased (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 3 | 4
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1
Graft versus host disease (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Anal infection (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 1 | 0
Ammonia increased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 7
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Coma (Nervous system disorders) | 1 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Thrombosis in device (Product Issues) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum1 Ph+ CP-CML; Dasatinib 60 mg/m^2 Starting Dose (N=17) | Stratum2/3 Ph+ALL or AP/BP-CML;Dasatinib60mg/m^2 Starting Dose (N=17) | Stratum4 Ph- ALL/AML; Dasatinib 60 mg/m^2 Starting Dose (N=24)
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 3
Palpitations (Cardiac disorders) | 3 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 2 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 3 | 0
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0 | 0
Chalazion (Eye disorders) | 1 | 0 | 0
Dacryoadenitis acquired (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Erythema of eyelid (Eye disorders) | 1 | 0 | 0
Eye discharge (Eye disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 2 | 0
Eye pruritus (Eye disorders) | 2 | 0 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 2
Eyelid ptosis (Eye disorders) | 0 | 1 | 0
Orbital oedema (Eye disorders) | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 1
Swelling of eyelid (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 9 | 2 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 11 | 7 | 6
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 6 | 13
Oral mucosal blistering (Gastrointestinal disorders) | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 9 | 7 | 11
Asthenia (General disorders) | 1 | 0 | 0
Catheter site erythema (General disorders) | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 2 | 2 | 0
Chills (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 7 | 4 | 4
Influenza like illness (General disorders) | 2 | 2 | 1
Injection site pain (General disorders) | 0 | 1 | 0
Injection site reaction (General disorders) | 1 | 1 | 0
Malaise (General disorders) | 3 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0
Pain (General disorders) | 3 | 3 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 5 | 8 | 8
Swelling (General disorders) | 1 | 0 | 0
Swelling face (General disorders) | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 2
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 2 | 1 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 1
Epididymitis (Infections and infestations) | 1 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0
Infection (Infections and infestations) | 2 | 1 | 2
Lice infestation (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 8 | 2 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 2 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 0
Rhinitis (Infections and infestations) | 3 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Viral rhinitis (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Body temperature (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 2 | 2
Heart rate increased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 4
Weight increased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Aneurysmal bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Epiphyses delayed fusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Growth retardation (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hypermobility syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 5 | 2
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 1
Facial paralysis (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 11 | 5 | 6
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Post-traumatic headache (Nervous system disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Enuresis (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Ovarian failure (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 5 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 6 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1 | 2
Flushing (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.